CLINICAL TRIAL: NCT05004831
Title: Phase II Study of Fruquintinib Combined With TAS-102 in the Treatment of Patients With Advanced Metastatic CRC
Brief Title: Fruquintinib Combined With TAS-102 in the Treatment of Patients With Advanced Metastatic CRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Peng Jian-jun, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C106
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib plus TAS-102 (Experimental): fruquintinib plus TAS-102, orally given, Q4W
  Interventions: Drug: fruquintinib plus TAS-102

INTERVENTIONS:
Drug: fruquintinib plus TAS-102 — fruquintinib 4mg/d, qd po, D1-21, Q4W; TAS-102 70mg/m2/d, bid po, D1-5, 8-12, Q4W

SUMMARY:
This phase II study aims to explore the efficacy and safety of fruquintinib combined with TAS-102 in the third-line treatment of patients with advanced metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a prospective, single center, one-arm phase II study. A total of 54 advanced mCRC patients refractory to standard therapies will be enrolled and administered with fruquintinib (4mg/d, qd po, D1-21, Q4W) combined with TAS-102 (70mg/m2/d, bid po, D1-5, 8-12, Q4W) until intolerable toxicity, disease progression or death. Primary endpoint of this study is PFS and secondary endpoints are OS, ORR, DCR and safety.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 75 years of age;
2. Histological or cytological confirmed advanced metastatic colorectal cancer;
3. Refractory to at least second line standard treatment containing fluorouracil, oxaliplatin and irinotecan;
4. At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan or 20mm by conventional CT scan);
5. ECOG performance status of 0-1;
6. Life expectancy ≥ 12 weeks;
7. No previous treatment with vascular endothelial growth factor receptor (VEGFR) inhibitor (TKI);
8. Signed and dated informed consent;
9. Adequate hepatic, renal, heart, and hematologic functions;
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Any factors that influence the usage of oral administration or any disease or condition that affects drug absorption;
3. Previous treatment with TAS-102;
4. Participated in clinical trials of other drugs within four weeks before enrollment;
5. Received other systemic anti-tumor therapy within 4 weeks before enrollment, including chemotherapy, signal transduction inhibitors, hormone therapy and immunotherapy;
6. International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN;
7. Clinically significant electrolyte abnormalities;
8. Subjected with hypertension that cannot be controlled by drugs, which is specified as: systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg;
9. Unrelieved toxic reactions higher than CTCAE V5.0 grade 1 caused by any previous anti-cancer treatment;
10. Incomplete healing of skin wound, surgical site, traumatic site, severe mucosal ulcer or fracture;
11. Conditions that may cause gastrointestinal bleeding and perforation determined by the researcher;
12. History of arterial thrombosis or deep venous thrombosis within 6 months before enrollment;
13. Stroke and / or transient cerebral ischemia occurred within 12 months before enrollment;
14. Cardiovascular diseases with significant clinical significance;
15. LVEF<50%;
16. Congestive heart failure New York Heart Association (NYHA) grade > 2;
17. Evidence of CNS metastasis;
18. Previous treatment with VEGFR inhibition;
19. Ventricular arrhythmias requiring drug treatment;
20. Proteinuria ≥ 2+ (1.0g/24hr);
21. Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy;
22. Other malignant tumors in the past 5 years, except skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
23. Active infection that is not controlled clinically, such as acute pneumonia, active hepatitis B or hepatitis C;
24. By judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
PFS | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  Progression-free Survival

SECONDARY OUTCOMES:
OS | from randomization until death due to any cause, assessed up to 3 years
  Overall Survival
DCR | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  Disease Control Rate
ORR | from randomization up to progressive disease or EOT due to any cause, up to 2 years
  Objective Response Rate
Safety and tolerance | from first dose to within 30 days after the last dose
  Safety and tolerance evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Peng, M.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China